## **Official Title:** The Feasibility of Using a Mobile Application for Training and Support of Elder Caregivers

**NCT:** NCT05877586

**IRB Document Date:** 7/12/2023

Verbal Consent for Digital Health Application for Training and Support of Elder Caregivers

**Interview Topic.** Based on your age and your loved one's age, you are eligible to participate in a pilot study on the use of technology in providing support and training to caregivers for home caregiving after hospital discharge of their loved ones. For this study, the technology that we will use is called CLARE, an application that is developed by the study's principal investigator, Dr. Cristina Hendrix. CLARE can be downloaded either to your smart phone or tablet. CLARE will contain materials on hospital discharge preparation, Covid care, and provide instructions on how to promote early mobility of your loved ones. CLARE will also help you use the After-Visit-Summary to determine home medications and information on follow-up appointments with patient's primary care providers. For you as a caregiver, CLARE will provide strategies on daily walking to promote your self-care. All information CLARE will provide comes from reliable sources including hospital documents. We will use CLARE to collect study data. You will have access to CLARE up to 7 days after hospital discharge. After 7 days of hospital discharge, your participation in the study will be complete. However, you may also be selected to participate in a 10-minute phone interview on your experience after you have used CLARE.

Potential Risks & Benefits. The potential small risk for this study includes loss of confidentiality; however, this is minimized by ensuring that all study data are stored in a secure server at Duke that only the study team can access. Also, if you are selected for the interview, we will encourage you not to mention your name or the name of your loved one (patient). The interview recording will also be stored on a secure server at Duke. We will not report individual data, rather, we will report data as a group. Pseudonyms will be used when we use your individual quotes in the interview for reporting. The direct benefit of participation in the study is additional support and training that you will receive as you provide care and assistance to your loved one after hospital discharge. The study may lead to information about the possibility of using an app to support caregivers after hospital discharge. Your participation will also contribute essential knowledge on how to modify CLARE to make it better and useful for caregivers.

Voluntary and Confidential Nature of Your Participation. Participating in this study is completely voluntary. The choice to do so is up to you. You are free to end participation at any time. Your responses will be kept completely confidential. We will do our best to make sure that information about you is kept confidential, but we cannot guarantee total confidentiality. Your personal information may be viewed by individuals involved in this research and may be seen by people including those collaborating, funding (i.e., NIH), and regulating the study. Also, by law, we will share with appropriate authorities any acts of child/elder abuse or domestic violence. Information about danger to yourself or others may also be shared to appropriate personnel such as your primary care provider. Data collected from you will only be used for purposes of this research. A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time. As a token of our appreciation for your time for participation, you will receive a gift card worth \$20.

DUHS IRB puestions. For questions about your rights as a research participant, or to discuss IRB NUMBER: Pro0111735
IRB REFERENCE DATE: 07/12/2023 suggestions related to the research, or to obtain information or IRB EXPRINTED TO THE EXPRINTED TO THE INSTITUTION OF THE EXPRINTED TO THE INSTITUTION OF THE INSTITUTION

| Review Board (IRB) Office at (919) 668-5111. If you have any questions about the study, you may contact the study team at (919) 684-9358. |
|---|
| Do you agree to the above information? |
| YesNo |
| ID Code # |

DUHS IRB IRB NUMBER: Pro00111735 IRB REFERENCE DATE: 07/

IRB REFERENCE DATE: 07/12/2023 IRB EXPIRATION DATE: 06/06/2025